CLINICAL TRIAL: NCT02395536
Title: Reveal LINQ™ In-Office 2 (RIO 2) Study United States
Brief Title: Medtronic Reveal LINQ™ In-Office 2 (RIO 2) Study United States
Acronym: RIO 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Version 1.0, 23 January 2015
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-05

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Masking Description: The site of the Reveal LINQ insertion was randomized. Therefore it was not possible to blind the subject or the investigator.
Oversight: Data Monitoring Committee: No

ARMS (2):
- In office Outside walls of hospital (Experimental): Reveal LINQ insertions will be performed in office setting. The in office setting was defined as a procedure or office room with controlled entry and hard floors outside the walls of the hospital and not an ambulatory surgery center.
  Interventions: Other: office setting
- Traditional Hospital Setting (Other): Reveal LINQ insertions will be performed in a traditional setting. The traditional hospital setting includes an operating room or electrophysiology laboratory.
  Interventions: Other: hosptial setting

INTERVENTIONS:
Other: office setting — An office setting was defined as a procedure or office room with controlled entry and hard floors outside the walls of the hospital and not including ambulatory surgical centers
  Arms: In office Outside walls of hospital
Other: hosptial setting — A hospital setting was defined as an operating room or electrophysiology lab inside the walls of a hospital.
  Arms: Traditional Hospital Setting

SUMMARY:
The primary purpose of the RIO 2 study is to demonstrate that when the Reveal LINQ™ insertable cardiac monitoring (ICM) system that records subcutaneous ECG insertion procedure performed in the in-office setting is as safe as LINQ™ insertions performed in the traditional hospital setting (operating room, cardiac catheterization or electrophysiology (EP) laboratory).

DETAILED DESCRIPTION:
RIO 2 is a two arm, randomized, prospective, un-blinded, multicenter, non-significant risk study. The primary objective for RIO 2 will be assessed by randomizing subjects to receive their LINQ™ insertion in the office setting or in the traditional hospital environment. Moving the LINQ™ insertion procedure to the office setting is not expected to decrease the complication rate compared to in hospital insertion procedures, however, moving the LINQ™ insertion procedure out of the traditional hospital setting may benefit the patient and reduce the burden to the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is indicated for continuous arrhythmia monitoring with a Reveal LINQ™ Insertable Cardiac Monitor
2. Patient is 18 years of age or older
3. Patient is willing to undergo ICM insertion procedure outside of the cath lab, OR, EP lab setting with only local anesthetic
4. Patient is willing and able to provide consent and authorize the use and disclosure of health information
5. Patient is willing and able to comply with the protocol including the required follow-up

Exclusion Criteria:

1. Patient has unusual thoracic anatomy or scarring at the implant site which may adversely affect the success of the implant procedure
2. Patient has reduced immune function or is otherwise at high risk for infection per physician discretion
3. Current therapy with immunosuppressive agents or chronic steroid use e.g. Prednisone greater than 20mg per day
4. Patient requires hemodialysis
5. Patient with active malignancy or history of chemotherapy or radiation treatment Patient has had a recent (within 30 days) or an active infection including but not limited to pneumonia, urinary tract, cellulitis, or bacteremia.
6. Patient has had major surgery (in the past 6 months)
7. Patient has undergone a procedure which required central venous or intraarterial access (e.g. AF/VT ablation, EP study, coronary angio) within the last 3 months or is scheduled for such a procedure while enrolled in the study.
8. Prior history of surgical infection, prosthetic device infection, or endovascular infection, including endocarditis, in the past 12 months.
9. Patient has a central venous port, an atrio-venous fistula, or a prosthetic valve
10. Patient requires conscious or moderate sedation to receive LINQ™
11. Patient is already implanted with a loop recorder
12. Patient is implanted or indicated for implant with a pacemaker, ICD, CRT device
13. Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager.
14. Patient's life expectancy is less than 6 months
15. Patient is pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Scripps Green Hospital, La Jolla, California
  - Saint Joseph Heritage Healthcare, Mission Viejo, California
  - Regional Cardiology Associates (Sacramento CA), Sacramento, California
  - Colorado Heart and Vascular, PC, Lakewood, Colorado
  - Cardiac Arrhythmia Service, Boca Raton, Florida
  - Clearwater Cardiovascular Consultants - Clearwater Office, Clearwater, Florida
  - Jim Moran Heart & Vascular-Holy Cross Hospital, Fort Lauderdale, Florida
  - Tallahassee Research Institute Inc, Tallahassee, Florida
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - Delmarva Heart Research Foundation Inc, Salisbury, Maryland
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Mid America Heart Institute (MAHI), Kansas City, Missouri
  - Lester E Cox Medical Center, Springfield, Missouri
  - Morristown Memorial Hospital, Newark, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Northwell Health, Great Neck, New York
  - The Mount Sinai Medical Center (New York NY), New York, New York
  - Cone Health Medical Group HeartCare at Church Street, Greensboro, North Carolina
  - Raleigh Cardiology Associates, Raleigh, North Carolina
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Diagnostic Cardiology Group, Chattanooga, Tennessee
  - Amarillo Heart Group, Amarillo, Texas
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Research Institute (Dallas TX), Dallas, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rogers JD, Piorkowski C, Sohail MR, Anand R, Kowalski M, Rosemas S, Stromberg K, Sanders P. Resource utilization associated with hospital and office-based insertion of a miniaturized insertable cardiac monitor: results from the RIO 2 randomized US study. J Med Econ. 2020 Jul;23(7):706-713. doi: 10.1080/13696998.2020.1746548. Epub 2020 May 1. PMID 32207636
- [Derived] Rogers JD, Sanders P, Piorkowski C, Sohail MR, Anand R, Crossen K, Khairallah FS, Kaplon RE, Stromberg K, Kowal RC. In-office insertion of a miniaturized insertable cardiac monitor: Results from the Reveal LINQ In-Office 2 randomized study. Heart Rhythm. 2017 Feb;14(2):218-224. doi: 10.1016/j.hrthm.2016.11.001. Epub 2016 Nov 4. PMID 27825975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 525 subjects were assessed for eligibility
Pre-assignment Details: 4 subjects excluded prior to randomization for not meeting inclusion/exclusion criteria
Groups:
- In Office Outside Walls of Hospital: Reveal LINQ insertions will be performed in office setting.
  Insertion of Reveal LINQ device in office or traditional hospital setting: The insterions will be performed in a Physician office setting or in Traditional Hospital Setting as per the arm the patient is randomized in.
- Traditional Hospital Setting: Reveal LINQ insertions will be performed in IN-a traditional setting
  Insertion of Reveal LINQ device in office or traditional hospital setting: The insterions will be performed in a Physician office setting or in Traditional Hospital Setting as per the arm the patient is randomized in.
Period: Overall Study
Arm/Group | In Office Outside Walls of Hospital | Traditional Hospital Setting
Started | 264 | 257
REVEAL LINQ Insertion (Number of subjects randomized that actually had a REVEAL LINQ insertion attempt) | 251 | 231
Completed | 244 | 227
Not Completed | 20 | 30
Not completed — Lost to Follow-up | 4 | 4
Not completed — Death | 2 | 0
Not completed — Physician Decision | 4 | 6
Not completed — Withdrawal by Subject | 9 | 17
Not completed — Inclusion/Excusion Criteria Violation | 1 | 2
Not completed — Insurance issue | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is the number of randomized subjects that had a REVEAL LINQ insertion attempt
Groups:
- Total: Total of all reporting groups
Arm/Group | In Office Outside Walls of Hospital | Traditional Hospital Setting | Total
Number analyzed (Participants) | 251 | 231 | 482
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (14.0) | 63.9 (14.9) | 64.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 125 | 242
  Male | 134 | 106 | 240
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 251 | 231 | 482
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (7.5) | 29.6 (7.1) | 30.0 (7.3)
Cardiomyopathy [Count of Participants; unit: Participants] | 9 | 8 | 17
Congestive heart failure [Count of Participants; unit: Participants] | 5 | 9 | 14
Hypertension [Count of Participants; unit: Participants] | 162 | 146 | 308
Myocardial infarction [Count of Participants; unit: Participants] | 13 | 10 | 23
Prior stroke or transient ischemic attack [Count of Participants; unit: Participants] | 69 | 58 | 127
Unexplained syncope [Count of Participants; unit: Participants] | 48 | 76 | 124
Paroxysmal atrial fibrillation [Count of Participants; unit: Participants] | 81 | 68 | 149
Persistent/permanent atrial fibrillation [Count of Participants; unit: Participants] | 14 | 14 | 28
Diabetes [Count of Participants; unit: Participants] | 43 | 53 | 96
Renal dysfunction [Count of Participants; unit: Participants] | 7 | 14 | 21

OUTCOME MEASURES:

1. Primary Outcome: Untoward Event Rate Associated With LINQ™ Insertions Performed
Description: Demonstrate that the untoward event rate associated with Reveal LINQ™ insertions performed in-office or in the traditional hospital setting (operating room, cardiac catheterization or EP laboratory) are comparable.
  Untoward events are a composite of unsuccessful Reveal LINQ™ or complications related to the Reveal LINQ™ insertion procedure or system.
Time Frame: 3 Months post insertion
Population: Subjects exiting prematurely (prior to 3-month visit) without an untoward event were excluded from primary analysis. There were 7 excluded from the In office arm (2 deaths unrelated to the REVEAL LINQ and 5 premature exits) and 4 excluded from the traditional hospital setting arm (all 4 due to premature exit)
Measure: Count of Participants; unit: Participants
Arm/Group | In Office Outside Walls of Hospital | Traditional Hospital Setting
Number analyzed (Participants) | 244 | 227
Participants | 2 | 2
Statistical Analysis 1: Comparison: In Office Outside Walls of Hospital vs Traditional Hospital Setting; The null hypothesis was that Reveal LINQ insertions performed in-office would have a higher untoward event rate than insertions performed in the traditional hospital setting. A sample size of 476 subjects was estimated to provide at least 90% power at a 1-sided alpha level of 2.5% and 5% non-inferiority margin. For the sample size calculation, an event rate of 2.0% was assumed in both arms. The Farrington-Manning test of two indepent proportions was used to compare study arms; Test type: Non-Inferiority — A non-inferiority margin of 5% was chosen since the inability to rule out a 5% increase in untoward event rate associated with moving the Reveal LINQ procedure in-office may suggest that in-office procedures would too high of a complication rate compared procedures performed in the traditional office setting; p < 0.001, Farrington-Manning test — P-value for non-inferiority versus a 5% non-inferiority margin; Risk Difference (RD) = -0.001, 95% CI 2-sided [-0.030 to 0.029] — The estimated value and its associated confidence interval are for the in-office minus traditional hospital setting difference in the untoward event rates. The point estimate is negative since the in-office rate was lower than the hospital rate

ADVERSE EVENTS:
Time Frame: All adeverse events potentially related to the REVEAL LINQ insertion procedure or system were collected from consent through the end of study participation (3-months post-procedure). Additionally all deaths were collected.
Description: An independent clinical events committee comprised on independent physicians who are not sponsor employees or study investigators and blinded to the subject's treatment arm adjudicated the relationship of each event to the REVEAL LINQ insertion procedure or system.
Arm/Group | In Office Outside Walls of Hospital | Traditional Hospital Setting
All-Cause Mortality (participants affected / at risk) | 2/251 | 0/231
Serious Adverse Events (participants affected / at risk) | 3/251 | 0/231
Other Adverse Events (participants affected / at risk) | 8/251 | 11/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Office Outside Walls of Hospital (N=251) | Traditional Hospital Setting (N=231)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Office Outside Walls of Hospital (N=251) | Traditional Hospital Setting (N=231)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 1 (1)
Device extrusion (General disorders) | 0 (0) | 1 (1)
Implant site bruising (General disorders) | 0 (0) | 1 (1)
Implant site rash (General disorders) | 0 (0) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Procedural dizziness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
It was not possible to blind either the subject or implanting physician. The study exit rate after randomization but prior to REVEAL LINQ procedure was relatively high, but not unexpected given randomization needed to occur prior to the procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes